CLINICAL TRIAL: NCT05801861
Title: Modulating Spatial Processing During Goal-directed Navigation Using Transcranial Magnetic Stimulation
Brief Title: Modulating Goal-directed Navigation Using Noninvasive Brain Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Travis Baker, PhD, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro2022000444_17-623R
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Spatial Navigation
Keywords: transcranial magnetic stimulation; spatial processing; EEG; neuroimaging
MeSH Terms: conditions — Spatial Navigation; Spatial Processing

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single (Participant) Participants will be blinded to the TMS condition (active or sham)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Active 10-Hz rTMS (Experimental): For the first TMS session, participants will receive 10-Hz repetitive TMS (rTMS) delivered at 110% of participants' resting motor threshold over the predefined parietal target for a total of 2250 pulses. For the second TMS session, participants will receive single pulse TMS during the phase target of each task trial and delivered at 110% of participants' resting motor threshold over the predefined parietal target for a total of 200 pulses.
  Interventions: Device: Active 10-Hz TMS to the parietal cortex
- Active single-pulse rTMS (Experimental): For the first TMS session, participants will receive a single TMS pulse during the phase target of each task trial and delivered at 110% of participants' resting motor threshold over the predefined parietal target for a total of 300 pulses. For the second TMS session, participants will receive single pulse TMS during the phase target of each task trial and delivered at 110% of participants' resting motor threshold over the predefined parietal target for a total of 200 pulses.
  Interventions: Device: Active single pulse TMS to the parietal cortex
- Sham 10-Hz rTMS (Sham Comparator): Identical parameters of the active 10-Hz rTMS group will be applied to the SHAM group with the exception that the TMS coil will be flipped 180º to mimic auditory stimulation.
  Interventions: Device: Sham 10-Hz TMS to the right parietal cortex
- Sham single-pulse rTMS (Sham Comparator): Identical parameters of the active single-pulse rTMS group will be applied to the SHAM group with the exception that the TMS coil will be flipped 180º to mimic auditory stimulation.
  Interventions: Device: Sham single-pulse rTMS the rigt parietal cortex

INTERVENTIONS:
Device: Active 10-Hz TMS to the parietal cortex — The active 10-Hz TMS group will receive 10hz TMS stimulation in the first TMS session, and single pulse TMS in the second TMS session. Participants in the active stimulation group will receive 10-Hz TMS to right parietal cortex. The TMS target will be based on subject specific anatomical MRI images (diffusion imaging). TMS will be delivered using a robotic neuronavigation system (Smartmove, ANT). Stimulation intensity will be standardized at 110% of RMT and adjusted to the skull to cortical surface based on e-field calculations (simnibs). Stimulation will be delivered to the right parietal cortex using an active/placebo figure-8 coil, an magventure TMS device.
  Arms: Active 10-Hz rTMS
Device: Active single pulse TMS to the parietal cortex — The active single pulse TMS group will receive single pulse TMS stimulation in the first and second TMS session. Participants in the active stimulation group will receive single pulse TMS to right parietal cortex. The TMS target will be based on subject specific anatomical MRI images (diffusion imaging). TMS will be delivered using a robotic neuronavigation system (Smartmove, ANT). Stimulation intensity will be standardized at 110% of RMT and adjusted to the skull to cortical surface based on e-field calculations (simnibs). Stimulation will be delivered to the right parietal cortex using an active/placebo figure-8 coil, an magventure TMS device.
  Arms: Active single-pulse rTMS
Device: Sham 10-Hz TMS to the right parietal cortex — The parameters in the active arms will be as above with the internal randomization of the device internally switching to sham in a blinded fashion.
  Arms: Sham 10-Hz rTMS
Device: Sham single-pulse rTMS the rigt parietal cortex — The parameters in the active arms will be as above with the internal randomization of the device internally switching to sham in a blinded fashion.
  Arms: Sham single-pulse rTMS

SUMMARY:
Our specific aim is to examine the effects of TMS on spatial processing during goal-directed navigation. In these experiments the investigators will utilize a scalp-recorded brain oscillation called right posterior theta that is believed to index the sensitivity of the parahippocampal cortex to spatial context. Here the investigators will asked whether this electrophysiological signal can be modulated up or down using TMS while participants engage in virtual navigation tasks, and if so, whether it would affect the spatial encoding of rewards and subsequent choices during task performance.

DETAILED DESCRIPTION:
The design is primarily a randomized control-trial design (3 sessions), testing the effects of 10-Hz rTMS and single-pulse TMS on spatial processing during goal-directed navigation tasks. Subjects will be randomly assigned to an active or sham group. All participants will be asked to complete two TMS sessions within two weeks. For the active TMS group, participants will be scanned using a 3 Tesla MRI system and will receive a structural (T1) and diffusion-weighted imaging (DWI) scan (Session A). For each subsequent TMS session, the TMS coil will be placed 1cm above the scalp over a right parietal region displaying maximum connectivity patterns with the parahippocampal cortex. Subjects will be randomly assigned to a 10-Hz rTMS protocol or single-pulse TMS protocol. At the start of the first TMS session (Session B), participants will be fitted with an EEG cap and engage in a virtual T-maze reward task. In this task, subjects will be asked to choose the left or right alley of the maze, and after their response, they will received a reward stimulus (apple or orange) which will indicate whether the participant will receive 5 or 0 cents on that trial. For the 10-Hz group, the task will be divided into 2 blocks (225 trials per block). At the start of Block 1, the robotic arm will position the TMS coil <1 cm over the right parietal target. Next, 50 rTMS pulses will be delivered at 110% of participants' rMT at 10-Hz continuously over the target immediately before every 10 trials of the T-maze. A total of 2250 pulses will be delivered and 450 T-maze trials completed. For the single-pulse group, the T-maze task will be divided into 2 blocks (225 trials per block). For the first block, a single TMS pulse will be delivered at 110% of participants' rMT over the TMS target immediately following trial-to-trial feedback and at the peak phase of the evoked theta oscillations (closed-loop). Following 10 trials of single-pulse, subjects will complete 5 trials with no TMS (total 150 TMS trials, 75 no-TMS trials). For the second block, a single TMS pulse will be delivered over the TMS target immediately following trial-to-trial feedback and at the trough phase of the evoked theta oscillation (peak and trough order will be counterbalanced across subjects). Following 10 trials of single-pulse, subjects will complete 5 trials with no TMS (total 150 TMS trials, 75 no-TMS trials). A total of 300 TMS trials and 150 no-TMS trials of the T-maze task will be performed. At the end of Session B, participants will be scheduled to return to the laboratory to complete Session C on a separate day. At the start of the second TMS session (Session C), participants will be fitted with an EEG cap and engage in the Linear Track Maze. During the encoding phase of this task, subjects will be presented with five distinct landmarks (pillars) along the track. Each time they reach a landmark, they stop for 500 ms and an apple (a reward, 5 cents) or an orange (no reward, 0 cents) appears. Only one landmark is associated with a reward. Following the encoding phase, the recall phase starts and subjects are shown both old and new landmarks. Subjects are instructed to indicate via button press which of these pillars was accompanied by a reward and earn the reward by correctly identifying the reward pillar. Recall performance will be assessed using d-prime, which represents how well subjects were able to recall the correct reward location. In total, subjects perform 200 trials across four blocks (50 trials each), resulting in a duration of roughly 30 minutes. For each block of the encoding phase, a single TMS pulses will be delivered at either at the peak, trough, ascending, descending phase of the evoked theta oscillation following the onset of the reward stimulus. (phase target order will be counterbalanced across blocks and subjects). The investigators will then test the effect of phase stimulation on recall performance as assed using d-prime. Identical protocols will be applied to the Sham groups with the exception that the TMS coil will be targeted at electrode position P4 and flipped 180 degrees, preventing pulses from hitting the scalp.

ELIGIBILITY:
Inclusion Criteria:

1. Be between the ages of 18 and 55 years old.
2. Not received substance abuse treatment within the previous 30 days.
3. Be in stable mental and physical health.
4. If female, test non-pregnant.
5. No evidence of focal or diffuse brain lesion on MRI.
6. Be willing to provide informed consent.
7. Be able to comply with protocol requirements and likely to complete all study procedures.

Exclusion Criteria:

1. Contraindication to MRI (e.g., presence of metal in the skull, orbits or intracranial cavity, claustrophobia).
2. Contraindication to rTMS (history of neurological disorder or seizure, increased intracranial pressure, brain surgery, or head trauma with loss of consciousness for > 15 minutes, implanted electronic device, metal in the head, or pregnancy).
3. History of autoimmune, endocrine, viral, or vascular disorder affecting the brain.
4. History or MRI evidence of neurological disorder that would lead to local or diffuse brain lesions or significant physical impairment.
5. Life time history of mental disorders such as: Bipolar Affective disorder (BPAD), Schizophrenia, Post-traumatic Stress disorder (PTSD) or Dementia or Major Depression.

uninterruptable central nervous system medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Event-related Brain Oscillation: Right Posterior Theta | Day 0 (day of testing)
  Right posterior theta (RPT: 4-8 hz) is a scalp recorded brain oscillation sensitive to spatial processing of reward stimulus presented during navigation tasks. RPT will be measured during the presentation of the reward stimulus (Reward, No-reward) during virtual navigation. A time-frequency analysis will be used to measure RPT power for each electrode by averaging the single-trial EEG according to feedback type (reward and no-reward) during the navigation tasks. The size of the RPT will be determined by identifying the maximum amplitude of the RPT response and evaluated at posterior electrodes. The RPT will be measured for each proposed right posterior target across active and sham groups, and used to measure the efficacy of the TMS target to modulate brain activity associated with spatial processing.
Spatial Recall performance | Day 0 (day of testing)
  Spatial recall performance learning will be measured using the Linear Track maze. During an initial encoding phase participants are exposed to five pairs of distinct pillars (landmarks), and only one of the pillar location will be paired with a reward cue. Then during the recall phase, participants are presented with old and new landmarks, and must recall which landmark contained the reward. A correct response would result in a 5-cent reward. Recall performance will be assessed using d-prime, which is calculated as the normalized distance between the probability distributions of the hit rate and the false alarm rate. This parameter represents how well subjects were able to maximize correct hits while minimizing false alarms. High recall performance is measured as a subject's ability to correctly identify rewarded pillars and reject non-rewarded pillars, as well as pillars that were not present during the last trial.

CONTACTS AND LOCATIONS:
Overall Officials: Travis E Baker, Principal Investigator — Rutgers University
Locations (1):
- Rutgers University - Newark, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Data may be uploaded to an open source framework. All data will be deidentified.